CLINICAL TRIAL: NCT02273024
Title: Exercise Therapy for Patients Awaiting Allogeneic Hematological Stem Cell Transplantation
Brief Title: Exercise Prior to Allogeneic Hematologic Stem Cell Transplantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other); Toronto Rehabilitation Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 14-7699
Record Dates: First submitted 2014-10-16; First posted 2014-10-23 (Estimated); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Allogeneic Stem Cell Transplantation
Keywords: Exercise; Quality of Life; Fatigue; Symptoms; Prehabilitation; Aerobic Capacity
MeSH Terms: conditions — Motor Activity; Fatigue | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Individuals will participate in weekly supervised and unsupervised exercise sessions prior to HSCT, during hospitalization and till 100 days from HSCT. Exercise will consist of endurance and resistance exercise 3-5 days a week.
  Interventions: Behavioral: Exercise
- Usual Care (No Intervention): Usual care will have continue with standard of care treatment without any specific exercise instruction or guidance other than what is provided by the patient education team at the cancer centre.

INTERVENTIONS:
Behavioral: Exercise
  Arms: Exercise

SUMMARY:
The investigators hypothesize that inactivity during the search for a donor may exacerbate current deconditioned states; subsequently, influencing risk factors for post-transplant complications that hinder the recovery phase.

This study is designed to investigate if exercise therapy administered prior to allogeneic hematologic stem cell transplantation (HSCT) can influence physical and psychological side-effects associated with HSCT. Approximately 6-weeks prior to HSCT, individuals will be randomized into either an exercise group or usual care group and followed until one year after HSCT.

ELIGIBILITY:
Inclusion Criteria:

* Medical indication: allogeneic stem cell transplantation at Princess Margaret Hospital
* must be ambulatory without need for human assistance at time of recruitment
* medically cleared to exercise by the transplant physician
* demonstrates willingness to attend supervised sessions
* sufficient in English to ensure safety of understanding prescribed exercise guidelines, or has access to an adequate non-familial interpreter

Exclusion Criteria:

* another active malignancy
* less than 4 weeks till the scheduled HSCT
* refusal to be randomized
* does not have the approval of their transplant physician
* severe or unstable neurological, cardiorespiratory, musculoskeletal disease or mental illness

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-10; Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Change in Physical Function | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  Cardiopulmonary Capacity (VO2peak)

SECONDARY OUTCOMES:
Change in Quality of Life | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  European Organization for Research and Treatment of Cancer (EORTC) core 30-item questionnaire (QLQ-30)
Change in Symptoms | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  Memorial Symptom Assessment Scale (MSAS)
Change in Anxiety | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  The Generalized Anxiety Disorder (GAD7)
Change in Depression | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  The Patient Health Questionnaire (PHQ-9), will be used as a clinically relevant measure to evaluate depression
Change in Fatigue | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  Multidimensional Fatigue Inventory
Change in Treatment Side-effects | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  Hospitalization (days till discharge and readmission rates), bone marrow engraftment (days), graft versus host disease incidence (acute & chronic), severity of diarrhea/ vomiting/ nausea, infections, steroid use, blood counts
Change in Strength | Baseline, 1 week pre HSCT, T100, 1yr post HSCT
  upper body: grip strength; lower body: chair-stand test
Change in Six-minute walk test | Baseline, 1 week pre HSCT, T100, 1yr post HSCT

OTHER OUTCOMES:
Adherence to exercise sessions | One year
  Feasibility of an exercise intervention prior to HSCT till T100

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Lipton, MD, PhD, Principal Investigator — Princess Margaret Hospital, University Health Network
Locations (1):
- Princess Margaret Hospital & Toronto Rehabilitation Institute, Toronto, Ontario, Canada